CLINICAL TRIAL: NCT02578550
Title: A Single-Dose, Open-Label, Randomized, Crossover Study to Assess the Bioequivalence of Darunavir 800 mg, Emtricitabine 200 mg, and Tenofovir Alafenamide 10 mg, in the Presence of Cobicistat 150 mg, Administered as Either a Fixed-Dose Combination Tablet or as Separate Agents in Healthy Subjects
Brief Title: A Bioequivalence Study of Darunavir, Emtricitabine, and Tenofovir Alafenamide, in the Presence of Cobicistat in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR107887; TMC114FD2HTX1001 (Other: Janssen Sciences Ireland UC); 2015-001264-18 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Immunodeficiency Virus Type 1, Human; Darunavir; Cobicistat; Emtricitabine; Tenofovir alafenamide; Healthy participants
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Cobicistat; emtricitabine tenofovir alafenamide; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence (AB) (Experimental): Participant will receive a single oral tablet of darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF fixed dose combination [FDC]) (Treatment A) in period 1, then 1 tablet of DRV 800 mg + 1 tablet of COBI 150 mg + 1 tablet of FTC/TAF 200/10 mg FDC (Treatment B) in period 2
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide fixed-dose combination (FDC); Drug: Emtricitabine/tenofovir alafenamide FDC; Drug: Darunavir; Drug: Cobicistat
- Treatment Sequence (BA) (Experimental): Participant will receive 1 tablet of DRV 800 mg + 1 tablet of COBI 150 mg + 1 tablet of FTC/TAF 200/10 mg FDC (Treatment B) in period 1, then a single oral tablet of D/C/F/TAF (800/150/200/10 mg) FDC (Treatment A) in period 2
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide fixed-dose combination (FDC); Drug: Emtricitabine/tenofovir alafenamide FDC; Drug: Darunavir; Drug: Cobicistat

INTERVENTIONS:
Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide fixed-dose combination (FDC) — A single tablet containing DRV 800 mg, COBI 150 mg, FTC 200 mg and TAF 10 mg will be administered.
Drug: Emtricitabine/tenofovir alafenamide FDC — A single tablet containing FTC 200 mg and TAF 10 mg will be administered.
Drug: Darunavir — A single tablet containing darunavir 800 mg will be administered.
Drug: Cobicistat — A single table containing cobistat 150 mg will be administered.

SUMMARY:
The purpose of this study is to evaluate the single-dose pharmacokinetics and pivotal bioequivalence of Darunavir (DRV) 800 milligram (mg), Emtricitabine (FTC) 200 mg, and tenofovir alafenamide (TAF) 10 mg when administered as a fixed-dose combination (FDC) (D/C/F/TAF) relative to the separate agents (DRV 800 mg tablet formulation and FTC/TAF 200/10 mg FDC) in the presence of 150 mg Cobicistat (COBI), under fed conditions, in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, 2-way crossover study in 96 healthy adult participants. The study consists of 2 treatment sessions. Participants will receive in one session a single dose of darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) 800/150/200/10 milligram (mg) tablets as fixed-dose combination (FDC) and in another session Darunavir (DRV) as 1x 800 mg tablet, Emtricitabine/ tenofovir alafenamide (FTC/TAF) as 1x 200/10 mg FDC tablet, and Cobicistat (COBI) 150 mg as 1x 150 mg tablet all under fed conditions. Treatment sessions will be separated by a washout period of at least 7 days. The duration of the study for an individual participant will be at least 12 days, Screening and Follow-up not included. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be non-smoker for at least 3 months prior to selection
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening. If the results are outside the normal reference ranges, the participant may be included only if they are not listed under the exclusion criteria and if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed/signed by the Investigator
* Participant must have a body mass index (BMI), between 18.5 and 30 kilogram per square meter (kg/m^2) (inclusive)
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening. If the results of the biochemistry panel, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the abnormalities or deviations from normal are not listed in the exclusion criteria, and the Investigator judges they are not clinically significant. This determination must be recorded in the participant's source documents and initialed/signed by the Investigator
* All female participants, except when postmenopausal, must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at Screening and must not breastfeed from Screening onwards

Exclusion Criteria:

* Participant has a positive human immunodeficiency virus - type (HIV-1) or human immunodeficiency virus - type 2 (HIV-2) test at Screening
* Participant has hepatitis A, B, or C infection (confirmed by a positive hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen, and/or hepatitis C virus antibody, respectively) at Screening
* Participant has currently significant and active gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, endocrinologic, genitourinary, renal, hepatic, respiratory, inflammatory, neoplastic, or infectious disease. Currently active dermatological disease that would interfere with a correct assessment of possible skin reactions to the study drugs
* Participant has currently significant and active diarrhea, nausea, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability
* Participant has any history of renal insufficiency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Darunavir, Cobicistat, Emtricitabine and Tenofovir Alafenamide | Up to 72 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Plasma Concentration at the Last Quantifiable Time Point (Clast) of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  The Clast is the last observed quantifiable plasma concentration above the quantification limit.
Elimination Rate Constant (Lambda[z]) of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  Lambda(z) is firstorder elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log linear phase of the drug concentrationtime curve.
Elimination HalfLife (t1/2) of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  The elimination halflife (t1/2) is the time needed for the plasma concentration to decrease to 1 half of its original value. It is associated with the terminal slope of the semi logarithmic drug concentrationtime curve, and is calculated as 0.693/lambda(z).
Time to Last Quantifiable Plasma Concentration (Tlast) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  The Tlast is the time to last observed quantifiable plasma concentration.
Ratio of AUClast of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  Ratio of individual AUClast values between Treatment A and B.
Ratio of AUC[0infinity] of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  Ratio of individual AUC[0infinity] values between Treatment A and B.
Ratio of Cmax of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 hours post-dose
  Ratio of individual Cmax values between Treatment A and B.
Number of Subjects with Adverse Events | From signing the Informed Consent Form (ICF) up to 10 days after last study drug administration
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Groningen, Netherlands

REFERENCES:
- [Derived] Crauwels HM, Baugh B, Van Landuyt E, Vanveggel S, Hijzen A, Opsomer M. Bioequivalence of the Once-Daily Single-Tablet Regimen of Darunavir, Cobicistat, Emtricitabine, and Tenofovir Alafenamide Compared to Combined Intake of the Separate Agents and the Effect of Food on Bioavailability. Clin Pharmacol Drug Dev. 2019 May;8(4):480-491. doi: 10.1002/cpdd.628. Epub 2018 Nov 9. PMID 30412360